CLINICAL TRIAL: NCT00137644
Title: Evaluation of the Preventing AIDS Through Live Movement and Sound (PALMS) Innovative HIV Prevention Intervention for Minority Adolescents by the Philadelphia Health Management Corporation in Philadelphia, PA
Brief Title: Evaluation of the Preventing AIDS Through Live Movement and Sound (PALMS) Intervention for Minority Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Public Health Management Corporation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-CCU324516; U65/CCU324516
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: Adolescent; *HIV Infections/ pc [Prevention & Control]; Male; Humans; Risk-Taking; Safe Sex; Sexual Behavior; HIV; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Risk-Taking; Safe Sex; Sexual Behavior | interventions — Sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Preventing AIDS Through Live Movement and Sound (PALMS)

SUMMARY:
The purpose of this program evaluation is to determine whether the Preventing AIDS Through Live Movement and Sound (PALMS) group-level intervention is effective in reducing HIV sex risk behaviors and increasing HIV testing of high-risk, incarcerated or adjudicated youth. The intent of this program is to support the evaluation of an existing intervention and provide feedback to the implementing organization for improved program effectiveness, not to conduct research.

DETAILED DESCRIPTION:
Philadelphia Health Management Corporation (PHMC) is evaluating the Preventing AIDS Through Live Movement and Sound (PALMS) group-level intervention for high-risk, incarcerated or adjudicated youth. PALMS uses three theater-based sessions to increase knowledge about HIV/AIDS, increase HIV testing, and reduce risky sexual behavior through increased self-efficacy. The intervention is delivered by peers, and peers work with the intervention team to use evaluation results to improve the program. The evaluation will recruit male adolescents, aged 12 to 18 years, who are residing in juvenile justice or drug treatment facilities in Philadelphia. The evaluation design uses concurrent intervention (N=132) and comparison (N=132) groups. Data will be collected at baseline, immediate post-intervention, and at a 6-month post-intervention follow-up. The intent of this program is to support the evaluation of an existing intervention and provide feedback to the implementing organization for improved program effectiveness, not to conduct research.

ELIGIBILITY:
Inclusion Criteria:

* Male adolescents
* Between the ages of 12 and 18
* Receiving residential services at juvenile justice or drug treatment facilities
* African-American or Latino

Exclusion Criteria:

* Do not speak English
* Prior participation in PALMS intervention
* Female adolescents

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 264 (Actual)
Dates: Start 2005-03; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Sexual activity | Within past 3 months & ever
Number and type (main and non-main) of female sex partners | Within past 3 months
Frequency of condom use with female sex partners | Within past 3 months
HIV testing (ever tested, number of tests, likelihood of test) | Within past 3 months

SECONDARY OUTCOMES:
Drug use | Within past 3 months
Knowledge of HIV transmission, prevention and testing | Concurrent
Attitudes and beliefs about condoms and safe sex | Concurrent
Beliefs about HIV and HIV testing | Concurrent
Perception of HIV risk | concurrent
Self-efficacy to use condoms and practice safe sex | Concurrent
Self-esteem | Concurrent
Perceptions of cultural and peer norms | Concurrent

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lauby, PhD, Principal Investigator — Public Health Management Corporation; Jeffrey H Herbst, PhD — Project Officer, Division of HIV/AIDS Prevention, NCHSTP, Centers for Disease Control and Prevention; Thomas M Painter, PhD — Project Officer, Division of HIV/AIDS Prevention, NCHSTP, Centers for Disease Control and Prevention
Locations (1):
- Philadelphia Health Management Corporation, Philadelphia, Pennsylvania, United States